CLINICAL TRIAL: NCT05389072
Title: Evaluation of The Comfort of Orthokeratology Lenses Fit Using A New Software
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CooperVision International Limited (CVIL) (Industry)
Collaborators: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEC-P042021
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Control Lens (Experimental)
  Interventions: Device: control contact lens

INTERVENTIONS:
Device: control contact lens — control CRT lens

SUMMARY:
As new orthokeratology fitting software emerges onto the market, it is of interest to assess their usefulness in guiding eye practitioners with lens fit. The goal of this study is to evaluate the comfort of Paragon orthokeratology lenses when they are fit using the new Procornea software.

ELIGIBILITY:
Inclusion Criteria:

1. Are 6- 35 years of age
2. Have had a self-reported visual exam in the last two years
3. Have a contact lens refraction that fits within the available parameters of the study lenses
4. Are able to read (or be read to), understand and sign the assent document if under 18 years old or are able to read, understand and sign the consent document if aged 18 or older (Children 6-years of age will not be asked to sign the assent form as per STERLING IRB.);
5. Are under 18 years old and are accompanied by a parent or legal guardian who is able to read, understand and sign the parental information and permission document;
6. Are willing to comply with the wear schedule (8 hour per night for every night, while sleeping)
7. Are willing to comply with the visit schedule
8. Have a refractive spherical component of their prescription between -0.50 and up to -6.00 diopters (inclusive) AND a refractive cylinder of no more than -1.75 diopters
9. Have a refractive spherical component ≥ cylinder component
10. Have a minimum visual acuity of +0.20 logMAR with each eye, when refracted at the Screening visit
11. Have clear corneas and no active ocular disease
12. Have no medication, medical condition, or ocular conditions that contraindicate contact wear OR are expected to affect lens comfort or vision across the 1-month study duration, in the opinion of the investigator
13. Can be shown to have stable keratometry for at least the previous 1 month, if they have previously worn orthokeratology lenses.

Exclusion Criteria:

1. Present at screening visit with the presence of ocular or systemic disease or reports the use medications which might interfere with orthokeratology contact lens wear, such as keratoconus, diabetes mellitus, steroid eye drops
2. Have a post-treatment predicted flat K value ≤38.00D (e.g. Patient baseline flat keratometry value = 40.00, patient has 2.00D of myopic refractive error. 40.00-2.00= 38.00D)
3. Have a known sensitivity to the diagnostic sodium fluorescein to be used in the study
4. Are pregnant, planning a pregnancy or lactating
5. Have amblyopia
6. Have presbyopia or has dependence on spectacles for near work over the contact lenses
7. Present at screening visit with the presence of clinically significant (grade >3; Efron scale) anterior segment abnormalities.
8. Present at screening visit with slit lamp findings that would contraindicate orthokeratology contact lens wear such as:

   1. Pathological dry eye or associated findings
   2. Pterygium, pinguecula, or corneal scars within the visual axis
   3. Neovascularization > 0.75 mm from of the limbus
   4. Giant papillary conjunctivitis (GPC) worse than grade 1
   5. Anterior uveitis or iritis (past or present)
   6. Seborrheic eczema, Seborrheic conjunctivitis
   7. History of corneal ulcers or fungal infections
   8. Poor personal hygiene
   9. Aphakia

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Comfort | 1 week
  Comfort of lenses (VAS 0-10, 0,5 steps) after insertion, subjects will be graded on a scale from 0 to 10 with 0=painful, 10= can't feel the lenses
Comfort | 1 month
  Comfort of lenses (VAS 0-10, 0,5 steps) after insertion, subjects will be graded on a scale from 0 to 10 with 0=painful, 10= can't feel the lenses

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - 4S Eyecare and Optometry, San Diego, California
  - Carillon Vision Care, Glenview, Illinois
  - Bellaire Family EyeCare, Bellaire, Texas
- University Complutense of Madrid, Madrid, Spain